CLINICAL TRIAL: NCT04218266
Title: Multicenter, Randomized, Active Comparator-controlled, Double-blind, Double-dummy, Parallel Group, Dose-finding Phase 2 Study to Compare the Safety of the Oral FXIa Inhibitor BAY2433334 to Apixaban in Patients With Atrial Fibrillation
Brief Title: Study to Gather Information About the Proper Dosing of the Oral FXIa Inhibitor BAY 2433334 and to Compare the Safety of the Study Drug to Apixaban, a Non-vitamin K Oral Anticoagulant (NOAC) in Patients With Irregular Heartbeat (Atrial Fibrillation) That Can Lead to Heart-related Complications.
Acronym: PACIFIC-AF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19765; 2019-002365-35 (EudraCT Number)
Record Dates: First submitted 2020-01-02; First posted 2020-01-06 (Actual); Results first posted 2022-10-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Atrial Fibrillation (AF)
MeSH Terms: conditions — Atrial Fibrillation | interventions — apixaban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BAY2433334 50mg+Apixaban matching placebo (Experimental)
  Interventions: Drug: BAY2433334; Other: Apixaban matching placebo
- BAY2433334 20mg+Apixaban matching placebo (Experimental)
  Interventions: Drug: BAY2433334; Other: Apixaban matching placebo
- BAY2433334 matching placebo+Apixaban (Active Comparator): Apixaban usual dose is 5 mg, reduced to 2.5 mg for participants with any 2 of the following criteria: age 80 years or older, body weight less than 60 kg, or serum creatinine level of 1.5 mg per dL or more.
  Interventions: Drug: Apixaban; Other: BAY2433334 matching placebo

INTERVENTIONS:
Drug: BAY2433334 — Tablet, taken orally once a day.
  Arms: BAY2433334 20mg+Apixaban matching placebo; BAY2433334 50mg+Apixaban matching placebo
Drug: Apixaban — Capsule, taken orally twice a day.
  Arms: BAY2433334 matching placebo+Apixaban
Other: BAY2433334 matching placebo — Tablet, taken orally once a day.
  Arms: BAY2433334 matching placebo+Apixaban
Other: Apixaban matching placebo — Capsule, taken orally twice a day.
  Arms: BAY2433334 20mg+Apixaban matching placebo; BAY2433334 50mg+Apixaban matching placebo

SUMMARY:
The purpose of this study is to try to find the best dose of the new drug BAY 2433334 to give to participants and to look at how well BAY 2433334 works in patients with irregular heartbeat (atrial fibrillation) that can lead to blood clots, stroke and other heart-related complications. In addition researchers want to compare the safety of the study drug to apixaban, a non-vitamin K oral anticoagulant (NOAC) in patients with atrial fibrillation. This study is also done to learn how the drug in this study moves into, through and out of the body. BAY 2433334, works by blocking a step of the blood clotting process in our body and thins the blood and is a so called oral FXIa inhibitor.

Apixaban, works by reducing the production of blood clotting factors in our body and thins the blood and is a so called non-vitamin K oral anticoagulant (NOAC). Thinning the blood can prevent you from blood clots which can cause a stroke.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 45 years of age or older at the time of signing the informed consent.
* Participant with AF documented by ECG evidence with

  * CHA2DS2-VASc score ≥ 2 if male or CHA2DS2-VASc score ≥ 3 if female
  * Indication for treatment with an oral anticoagulant in

    * any participant currently not treated with an oral anticoagulant (e.g. treatment naïve) or alternatively,
    * participant on a NOAC in case of at least one bleeding risk feature (history of a prior bleed within the last 12 months requiring medical attention and / or moderate renal dysfunction with eGFR 30-50 ml/min and / or current clinically indicated antiplatelet therapy with Acetylsalicylic acid(ASA) ≤ 100 mg)
* Written informed consent

Exclusion Criteria:

* Mechanical heart valve prosthesis
* Any degree of rheumatic mitral stenosis or moderate-to-severe, non-rheumatic mitral stenosis
* Atrial fibrillation due to a reversible cause, participants in sinus rhythm after successful ablation, or plan for cardioversion or ablation during study conduct
* Requirement for chronic anticoagulation (for a different indication than AF) or antiplatelet therapy (up to 100 mg ASA is allowed). Anticipated need for chronic therapy with Nonsteroidal anti-inflammatory drugs (NSAIDs)
* Treated with a Vitamin K antagonist in the 30 days prior to screening

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 755 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2021-10-08 (Actual); Study Completion 2021-10-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (92):
- Austria (8):
  - Medizinische Universität Graz, Graz, Styria
  - Medizinische Universität Innsbruck, Innsbruck, Tyrol
  - Krankenhaus St. Josef Braunau, Braunau am Inn, Upper Austria
  - Ordensklinikum Linz GmbH Elisabethinen, Linz, Upper Austria
  - Landeskrankenhaus Feldkirch, Feldkirch, Vorarlberg
  - Uniklinikum Salzburg - Landeskrankenhaus, Salzburg
  - Universitätsklinikum AKH Wien, Vienna
  - Klinik Floridsdorf - Krankenhaus Nord, Vienna
- Belgium (7):
  - UZ Leuven Gasthuisberg, Leuven, Vlaams Brabant
  - Imeldaziekenhuis - St-Elisabethkliniek, Bonheiden
  - AZ St-Jan Brugge Oostende AV, Bruges
  - UZ Antwerpen, Edegem
  - Jessa Ziekenhuis, Hasselt
  - VZW Emmaus, Mechelen
  - AZ Delta, Roeselare
- Canada (4):
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Montreal Heart Institute, Montreal, Quebec
  - Clinique Sante Cardio MC, Montreal, Quebec
  - Institut universitaire de cardiologie et de pneumologie, Ste-Foy, Quebec
- Czechia (6):
  - Fakultni nemocnice Plzen - Lochotin, Pilsen
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Institut Klinicke a Experimentalni Mediciny, Prague
  - Fakultni nemocnice v Motole, Prague
  - Nemocnice Slany, Slaný
  - Krajska nemocnice T. Bati, a.s., Zlín
- France (7):
  - Hôpital Henri Mondor, Créteil
  - Centre Hospitalier Départemental Vendée, La Roche-sur-Yon
  - Centre Hospitalier Louis Pasteur, Le Coudray
  - Hopital Bichat - Paris, Paris
  - Centre Hospitalier Régional - Saint Brieuc, Saint-Brieuc
  - Hôpital de Rangueil - Toulouse, Toulouse
  - Centre Hospitalier - Valenciennes Cedex, Valenciennes
- Hungary (8):
  - Tagore Medical Center, Balatonfüred
  - University of Semmelweis/ Semmelweis Egyetem, Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - Kanizsai Dorottya Hospital, Nagykanizsa
  - Medifarma-98 Egeszsegugyi, Kereskedelmi es Szolgaltato Kft., Nyíregyháza
  - Pecsi Tudomanyegyetem Klinikai Kozpont, Pécs
  - Tolna Megyei Balassa Janos Korhaz, Szekszárd
  - Csongrad-Csanad Megyei Dr. Bugyi Istvan Korhaz, Szentes
- Italy (6):
  - A.O.U. Policlinico Umberto I, Rome, Lazio
  - IRCCS Ospedale Policlinico San Martino, Genoa, Liguria
  - ASST Spedali Civili di Brescia, Brescia, Lombardy
  - ASUR Marche - Area Vasta 5, Ascoli Piceno, The Marches
  - AUSL Toscana Sud-Est, Arezzo, Tuscany
  - A.O. di Perugia, Perugia, Umbria
- Japan (9):
  - Nakamura Cardiovascular Clinic, Itoshima, Fukuoka
  - Hyogo Prefectural Harima-Himeji General Medical Center, Himeji, Hyōgo
  - Hayama Heart Center, Miura-gun, Kanagawa
  - Kishiwada Tokushukai Hospital, Kishiwada, Osaka
  - Yao Tokushukai General Hospital, Yao, Osaka
  - Nishiarai Heart Central Clinic, Adachi-ku, Tokyo
  - Minamino Cardiovascular Hospital, Hachiōji, Tokyo
  - Tokyo Angel Hospital, Hachiōji, Tokyo
  - Koto Hospital, Koto-ku, Tokyo
- Latvia (6):
  - Doctor's Practice in Cardiology, Daugavpils
  - Daugavpils Regional Hospital, Daugavpils
  - Liepaja Regional Hospital, Liepāja
  - 1st Riga Clinical Hospital, Riga
  - P. Stradins Clinical University Hospital, Riga
  - Riga East Clinical University Hospital "Gailezers", Riga
- Netherlands (8):
  - Academisch Medisch Centrum (AMC), Amsterdam
  - Ziekenhuis Rijnstate, Arnhem
  - Amphia Ziekenhuis, locatie Molengracht, Breda
  - Albert Schweitzer Ziekenhuis, Dordwijk, Dordrecht
  - Medisch Spectrum Twente, Enschede
  - Martini Ziekenhuis, Locatie van Swieten, Groningen
  - Spaarne Gasthuis - locatie Zuid, Haarlem
  - Maastricht UMC, Maastricht
- Spain (5):
  - Ciutat Sanitària i Universitària de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Ciutat Sanitària i Universitaria de la Vall d'Hebron, Barcelona
  - Hospital de la Santa Creu i de Sant Pau | Cardiología, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Virgen de la Victoria, Málaga
- Sweden (7):
  - Falu Lasarett, Falun
  - Clemenstorget Hjärtmottagning, Lund
  - Avdelningen för kliniska prövningar AKP, Örebro
  - Östersunds Sjukhus, Östersund
  - Skellefteå Lasarett, Skellefteå
  - Södersjukhuset AB, Stockholm
  - Danderyds sjukhus, Stockholm
- Switzerland (6):
  - Kantonsspital Aarau, Aarau, Canton of Aargau
  - Universitätsspital Basel, Basel, Canton of Basel-City
  - Kantonsspital St. Gallen, Sankt Gallen, Canton of St. Gallen
  - Inselspital Universitätsspital Bern, Bern
  - Hôpital Cantonal Universitaire de Genève, Geneva
  - Ospedale regionale di Lugano, Lugano
- United Kingdom (5):
  - Staploe Medical Centre, Ely, Cambridgeshire
  - Queen Elizabeth II Hospital, Welwyn Garden City, Hertfordshire
  - Northwick Park Hospital, Harrow, London
  - St Richard's Hospital, Chichester, West Sussex
  - Heart and Chest Hospital, Liverpool

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Derived] Piccini JP, Caso V, Connolly SJ, Fox KAA, Oldgren J, Jones WS, Gorog DA, Durdil V, Viethen T, Neumann C, Mundl H, Patel MR; PACIFIC-AF Investigators. Safety of the oral factor XIa inhibitor asundexian compared with apixaban in patients with atrial fibrillation (PACIFIC-AF): a multicentre, randomised, double-blind, double-dummy, dose-finding phase 2 study. Lancet. 2022 Apr 9;399(10333):1383-1390. doi: 10.1016/S0140-6736(22)00456-1. Epub 2022 Apr 3. PMID 35385695
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field. — http://clinicaltrials.bayer.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 94 centers in 14 countries or regions, between 30-Jan-2020 (first participant first visit) and 08-Oct-2021 (last participant last visit)
Pre-assignment Details: 862 participants were screened. 107 participants were screening failures. 755 participants were randomized in a 1:1:1 ratio to 3 treatment groups: 251 participants to the asundexian 20 mg group, 254 participants to the asundexian 50 mg group and 250 participants to the apixaban group. 2 participants of asundexian 20 mg group never administered drug.
Groups:
- Asundexian 20 mg: Participants received Asundexian (BAY2433334) 20 mg and Apixaban placebo for 12 weeks
- Asundexian 50 mg: Participants received Asundexian (BAY2433334) 50 mg and Apixaban placebo for 12 weeks
- Apixaban: Participants received Asundexian (BAY2433334) placebo and Apixaban for 12 weeks
Period: Overall Study
Arm/Group | Asundexian 20 mg | Asundexian 50 mg | Apixaban
Started (Randomized) | 251 | 254 | 250
Treated | 249 | 254 | 250
Completed | 226 (Treatment completed) | 227 (Treatment completed) | 218 (Treatment completed)
Not Completed | 25 | 27 | 32
Not completed — Death | 1 | 2 | 3
Not completed — Adverse Event | 13 | 14 | 11
Not completed — Other | 7 | 5 | 14
Not completed — Physician Decision | 1 | 3 | 2
Not completed — Non-compliance with study drug | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 3 | 1
Not completed — Study drug never administered | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: SAF (safety analysis set)
Groups:
- Total: Total of all reporting groups
Arm/Group | Asundexian 20 mg | Asundexian 50 mg | Apixaban | Total
Number analyzed (Participants) | 249 | 254 | 250 | 753
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 33 | 43 | 34 | 110
  >=65 years | 216 | 211 | 216 | 643
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 97 | 109 | 308
  Male | 147 | 157 | 141 | 445
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 39 | 40 | 40 | 119
  Black or African American | 1 | 1 | 1 | 3
  White | 209 | 212 | 209 | 630
  Not reported | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants With All Bleeding
Description: Adjudication of all bleeding events was performed by members of the Clinical events committee (CEC) who reviewed events in a blinded fashion and adjudicated and classified the following events in a consistent and unbiased manner according to the following classifications: ISTH (major, clinically relevant non-major and minor); Thrombolysis in myocardial infarction (TIMI major, minor, requiring medical attention, minimal); Bleeding Academic Research Consortium (BARC type 1, 2, 3, 5).
Time Frame: After the first administration of study intervention with an average administration of 12 weeks (but not starting after more than 2 days after the last administration)
Population: Safety analysis set (SAF)
Measure: Count of Participants; unit: Participants
Groups:
- Asundexian Pooled: Asundexian 20 mg group and Asundexian 50 mg group
Arm/Group | Asundexian 20 mg | Asundexian 50 mg | Asundexian Pooled | Apixaban
Number analyzed (Participants) | 249 | 254 | 503 | 250
Participants | 12 | 10 | 22 | 26
Statistical Analysis 1: Comparison: Asundexian Pooled vs Apixaban; Comparison of the Asundexian pooled group (Asundexian 20 mg group and Asundexian 50 mg group) versus Apixaban group in all bleeding; Test type: Other; Crude incidence ratio = 0.42, 90% CI 2-sided [0.26 to 0.67]

2. Secondary Outcome: Number of Participants With ISTH Major Bleeding
Description: ISTH Major Bleeding criteria: 1. Fatal bleeding, and/or 2. Symptomatic bleeding in a critical area or organ (intracranial, intraocular, intraspinal, pericardial, retroperitoneal, intraarticular, or intramuscular with compartment syndrome), and/or 3. Clinically overt bleeding associated with a recent decrease in the hemoglobin level of ≥ 2 g/dL (20 g/L; 1.24 mmol/L) compared to the most recent hemoglobin value available before the event, and/or 4. Clinically overt bleeding leading to transfusion of 2 or more units of packed red blood cells or whole blood.
Time Frame: as for outcome 1
Population: Safety analysis set (SAF)
Measure: Count of Participants; unit: Participants
Arm/Group | Asundexian 20 mg | Asundexian 50 mg | Apixaban
Number analyzed (Participants) | 249 | 254 | 250
Participants | 0 | 0 | 0

3. Secondary Outcome: Number of Participants of ISTH Clinically Relevant Non-major (CRNM) Bleeding
Description: ISTH Clinically Relevant Non-Major Bleeding is considered any sign or symptom of hemorrhage that does not fit the criteria for the ISTH definition of major bleeding, but does meet at least one of the following criteria 1. requiring medical intervention by a healthcare professional. 2. leading to hospitalization or increased level of care. 3. prompting a face to face (i.e. not just a telephone or electronic communication) evaluation.
Time Frame: as for outcome 1
Population: Safety analysis set (SAF)
Measure: Count of Participants; unit: Participants
Arm/Group | Asundexian 20 mg | Asundexian 50 mg | Asundexian Pooled | Apixaban
Number analyzed (Participants) | 249 | 254 | 503 | 250
Participants | 3 | 1 | 4 | 6
Statistical Analysis 1: Comparison: Asundexian Pooled vs Apixaban; Comparison of the Asundexian pooled group (Asundexian 20 mg group and Asundexian 50 mg group) versus Apixaban group in ISTH CRNM bleeding; Test type: Other; Crude incidence ratio = 0.33, 90% CI 2-sided [0.09 to 0.97]

4. Secondary Outcome: Number of Participants With ISTH Minor Bleeding
Description: All other overt bleeding episodes not meeting ISTH Major Bleeding criteria or clinically relevant non major bleeding were classified as minor bleeding.
Time Frame: as for outcome 1
Population: Safety analysis set (SAF)
Measure: Count of Participants; unit: Participants
Arm/Group | Asundexian 20 mg | Asundexian 50 mg | Asundexian Pooled | Apixaban
Number analyzed (Participants) | 249 | 254 | 503 | 250
Participants | 10 | 9 | 19 | 20
Statistical Analysis 1: Comparison: Asundexian Pooled vs Apixaban; Comparison of the Asundexian pooled group (Asundexian 20 mg group and Asundexian 50 mg group) versus Apixaban group in ISTH minor bleeding; Test type: Other; Crude incidence ratio = 0.47, 90% CI 2-sided [0.28 to 0.83]

5. Primary Outcome: Number of Participants With Composite of International Society on Thrombosis and Hemostasis (ISTH) Major Bleeding or Clinically Relevant Non-major (CRNM) Bleeding
Description: ISTH Major Bleeding criteria: 1. Fatal bleeding, and/or 2. Symptomatic bleeding in a critical area or organ (intracranial, intraocular, intraspinal, pericardial, retroperitoneal, intraarticular, or intramuscular with compartment syndrome), and/or 3. Clinically overt bleeding associated with a recent decrease in the hemoglobin level of ≥ 2 g/dL (20 g/L; 1.24 mmol/L) compared to the most recent hemoglobin value available before the event, and/or 4. Clinically overt bleeding leading to transfusion of 2 or more units of packed red blood cells or whole blood.
  ISTH Clinically Relevant Non-Major Bleeding is considered any sign or symptom of hemorrhage that does not fit the criteria for the ISTH definition of major bleeding, but does meet at least one of the following criteria 1. requiring medical intervention by a healthcare professional. 2. leading to hospitalization or increased level of care. 3. prompting a face to face (i.e. not just a telephone or electronic communication) evaluation.
Time Frame: as for outcome 1
Population: Safety analysis set (SAF)
Measure: Count of Participants; unit: Participants
Arm/Group | Asundexian 20 mg | Asundexian 50 mg | Asundexian Pooled | Apixaban
Number analyzed (Participants) | 249 | 254 | 503 | 250
Participants | 3 | 1 | 4 | 6
Statistical Analysis 1: Comparison: Asundexian Pooled vs Apixaban; Comparison of the Asundexian pooled group (Asundexian 20 mg group and Asundexian 50 mg group) versus Apixaban group in ISTH major bleeding or CRNM bleeding; Test type: Other; Other; Crude incidence ratio = 0.33, 90% CI 2-sided [0.09 to 0.97]

ADVERSE EVENTS:
Time Frame: After the first administration of study intervention with an average administration of 12 weeks (but not starting after more than 2 days after the last administration). Adverse event reporting for the all-cause mortality considers all deaths that occurred at any time during the study before the last contact, with an average of 14 weeks.
Arm/Group | Asundexian 50 mg | Asundexian 20 mg | Apixaban
All-Cause Mortality (participants affected / at risk) | 4/254 | 2/249 | 5/250
Serious Adverse Events (participants affected / at risk) | 20/254 | 22/249 | 20/250
Other Adverse Events (participants affected / at risk) | 116/254 | 110/249 | 113/250
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asundexian 50 mg (N=254) | Asundexian 20 mg (N=249) | Apixaban (N=250)
Atrial fibrillation (Cardiac disorders) | 3 (4) | 3 (3) | 2 (2)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Cardiac failure (Cardiac disorders) | 4 (4) | 3 (4) | 3 (3)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial thrombosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Congestive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Face oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Sudden cardiac death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Cardiac ablation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Percutaneous coronary intervention (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asundexian 50 mg (N=254) | Asundexian 20 mg (N=249) | Apixaban (N=250)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0)
Polycythaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Spontaneous haematoma (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 2 (2) | 2 (2) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 8 (9) | 7 (7) | 7 (7)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 1 (2)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
Cardiac failure (Cardiac disorders) | 0 (0) | 2 (2) | 5 (5)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
Cardiomegaly (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 4 (4) | 3 (3) | 1 (2)
Sinus bradycardia (Cardiac disorders) | 3 (3) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Accessory spleen (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 4 (4) | 2 (2) | 3 (3)
Vertigo labyrinthine (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 2 (2)
Autoimmune thyroiditis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 2 (2) | 2 (2)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Myopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Swelling of eyelid (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 2 (2)
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 2 (2) | 6 (6)
Change of bowel habit (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 11 (11) | 4 (5) | 5 (5)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 3 (3) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (8) | 6 (7) | 9 (10)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oral discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Saliva altered (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1)
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal symptom (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 3 (3) | 4 (4)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 2 (2) | 3 (3) | 0 (0)
Discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 10 (10) | 5 (5) | 2 (2)
Feeling abnormal (General disorders) | 1 (1) | 1 (1) | 0 (0)
Feeling cold (General disorders) | 3 (3) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 1 (1)
Oedema (General disorders) | 1 (1) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 3 (3) | 2 (2) | 3 (3)
Pain (General disorders) | 2 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Thirst (General disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 1 (1)
Hernia pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0)
Inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 1 (1) | 0 (0)
Medical device site inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic fibrosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Amyloidosis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3) | 1 (1) | 2 (3)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Pulpitis dental (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tinea cruris (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 3 (3)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gingival abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oral fungal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Haematuria traumatic (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 3 (3)
Inflammation of wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skin wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 3 (3)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Heart rate decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Reticulocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight increased (Investigations) | 0 (0) | 2 (2) | 1 (1)
Urinary occult blood positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Angiocardiogram (Investigations) | 1 (1) | 0 (0) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Folate deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (5) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 8 (8) | 9 (9) | 7 (10)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Essential tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Head discomfort (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 7 (7) | 4 (4) | 5 (5)
Hypertonia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Neuritis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0)
Parkinsonism (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Orthostatic intolerance (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (3) | 1 (1) | 1 (1)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 6 (6)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 3 (3) | 2 (2) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 3 (3) | 3 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (8) | 3 (3) | 11 (12)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pharyngeal paraesthesia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Intertrigo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (5) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Cardioversion (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Cataract operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 3 (3)
Hypertension (Vascular disorders) | 5 (6) | 6 (6) | 7 (7)
Hypotension (Vascular disorders) | 1 (1) | 2 (2) | 3 (3)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral coldness (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Phlebitis superficial (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Subclavian artery thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertensive urgency (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-09-25): https://cdn.clinicaltrials.gov/large-docs/66/NCT04218266/Prot_002.pdf
  • Statistical Analysis Plan (2021-10-14): https://cdn.clinicaltrials.gov/large-docs/66/NCT04218266/SAP_003.pdf